CLINICAL TRIAL: NCT06541678
Title: A Phase 1, Open-Label, Fixed-Sequence Study to Evaluate the Effect of Itraconazole and Cyclosporine on the Single-Dose Pharmacokinetics of Danuglipron in Healthy Adult Participants
Brief Title: A Study to Learn if the Study Medicines Called Itraconazole and Cyclosporine Change How the Body Processes the Other Study Medicine Called Danuglipron in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3421063; 2024-513863-21-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: danuglipron; cyclosporine; itraconazole; DDI
MeSH Terms: interventions — danuglipron; Cyclosporine; Itraconazole

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, open-label, fixed-sequence, 3-period study
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Period 1: Danuglipron (Active Comparator): Participants will receive a single 20 mg dose of danuglipron on Day 1.
  Interventions: Drug: Danuglipron
- Period 2: Cyclosporine + Danuglipron (Experimental): Participants will receive a single 20 mg dose of danuglipron and a single 600 mg dose of cyclosporine on Day 1.
  Interventions: Drug: Danuglipron; Drug: Cyclosporine
- Period 3: Itraconazole + Danuglipron (Experimental): Participants will receive itraconazole daily for 6 days plus a single dose of danuglipron on Day 4.
  Interventions: Drug: Danuglipron; Drug: Itraconazole

INTERVENTIONS:
Drug: Danuglipron — MR Tablet
  Other Names: PF-06882961
Drug: Cyclosporine — Capsule
  Arms: Period 2: Cyclosporine + Danuglipron
Drug: Itraconazole — Oral solution
  Arms: Period 3: Itraconazole + Danuglipron

SUMMARY:
The purpose of this study is to see how single dose of cyclosporine and multiple doses of itraconazole affect the level of the study medicine danuglipron in the blood of healthy adult participants. The information from this study may inform how danuglipron will be used in the future with medicines like cyclosporine and itraconazole.

DETAILED DESCRIPTION:
This study is seeking healthy participants who:

* are aged 18 years of age or older.
* are confirmed to be healthy by some medical tests.
* both men and women can participate. Women who can produce a baby must agree to use a highly effective method of birth control.
* have body mass index (BMI) of 16 to 32 kilograms per meter squared.
* a total body weight of more than 50 kilograms.

Participants will receive danuglipron tablet by mouth on Day 1. Then on Day 4, participants will take cyclosporine capsules and danuglipron tablet by mouth at the same time. From Day 7 of the study, participants will take itraconazole solution by mouth once a day until Day 12. On Day 10 of the study, danuglipron tablet will also be taken with itraconazole at the same time.

The total planned time of participation is about 10 weeks. The study consists of:

screening period of up to 28 days before taking sisunatovir. 13 days of staying in the study clinic. a follow-up contact that will occur 28 to 35 days after taking itraconazole the last time.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female 18 years of age or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, blood pressure, pulse rate and standard 12-lead ECG.
2. BMI of 16-32 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal (including acute pancreatitis or a history of chronic pancreatitis), cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
   * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
   * Known intolerance or hypersensitivity to GLP-1R agonists.
   * Known hypersensitivity to itraconazole or cyclosporine.
2. Personal or family history of MTC or MEN2, or participants with suspected MTC per the investigator's judgment.
3. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
4. Use of prescription or nonprescription drugs and dietary and herbal supplements within 14 days or 5 half lives (whichever is longer; 14 days plus 5 half-lives for moderate or strong CYP3A inducers) prior to the first dose of study intervention (Refer to Section 6.9 for additional details).
5. Prior or current use of any prohibited concomitant medication(s) (Refer to Section 6.9 for additional details).

   Prior/Concurrent Clinical Study Experience:
6. Previous administration of an investigational product (drug or vaccine) within 30 days or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.
7. Known prior participation (ie, randomized and received at least 1 dose of investigational product) in a study involving danuglipron.
8. A positive urine drug test at Screening or Day -1.
9. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥140 or 150 mm Hg (based on age) or diastolic BP ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
10. An eGFR (<60 units of mL/min/1.73 m²) as determined by the CKD-EPI equation using Screat as described in Section 10.7.2.
11. Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST segment and/or T wave changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer interpreted ECGs should be overread by an investigator experienced in reading ECGs before excluding a participant.
12. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * ALT or AST ≥1.5× ULN;
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ULN;
    * Hemoglobin A1c (HbA1c) ≥6.5%;
    * Fasting blood glucose ≥126 mg/dL (7 mmol/L).
13. History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence within 6 months of screening.
14. Use of tobacco/nicotine containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
AUCinf (if data permits otherwise AUClast): to estimate the effect of a single dose of cyclosporine on the single-dose PK of a MR formulation of danuglipron in healthy adult participants. | 0 to 72 hour postdose
  AUCinf: Area under the plasma concentration time profile from time zero extrapolated to infinite time
  AUClast: Area under the plasma concentration time profile from time zero to the time of the last quantifiable concentration.
Cmax: to estimate the effect of a single dose of cyclosporine on the single-dose PK of a MR formulation of danuglipron in healthy adult participants. | 0 to 72 hour postdose
  Maximum observed plasma concentration
AUCinf (if data permits otherwise AUClast): to estimate the effect of multiple doses of itraconazole on the single-dose PK of a MR formulation of danuglipron in healthy adult participants. | 0 to 72 hour postdose
  AUCinf: Area under the plasma concentration time profile from time zero extrapolated to infinite time
  AUClast: Area under the plasma concentration time profile from time zero to the time of the last quantifiable concentration.
Cmax: to estimate the effect of multiple doses of itraconazole on the single-dose PK of a MR formulation of danuglipron in healthy adult participants. | 0 to 72 hour postdose
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events Following Single Doses of Danuglipron administered separately and in combination with itraconazole or cyclosporine | Day 1 up to approximately Day 47
Number of Participants With Clinical Laboratory Abnormalities Following Single Doses of Danuglipron administered separately and in combination with itraconazole or cyclosporine | Day 1 up to approximately Day 47
Number of Participants With Clinically Significant Change from Baseline Vital Signs Following Single Doses of Danuglipron administered separately and in combination with itraconazole or cyclosporine | Day 1 up to approximately Day 47
Number of Participants With Clinically Significant Change from Baseline in Electrocardiogram Findings Following Single Doses of Danuglipron administered separately and in combination with itraconazole or cyclosporine | Day 1 up to approximately Day 47

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421063